CLINICAL TRIAL: NCT02023086
Title: Clinical Investigation on the Blood Oxygenation at the Optic Nerve Head in Relation With Visual Field Loss in Fabry Patients
Brief Title: Clinical Investigation on the Blood Oxygenation at the Optic Nerve Head in Fabry Patients
Status: Completed | Type: Observational
Sponsor: Université de Montréal (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Langis Michaud, Professor, Université de Montréal
Other Study IDs: GZ-2012-10918
Record Dates: First submitted 2013-12-10; First posted 2013-12-30 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fabry Disease
Keywords: Visual field defect; Blood oxygenation; Optic nerve Head
MeSH Terms: conditions — Fabry Disease | interventions — Visual Fields; Tropicamide; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FABRY group: * contrast sensitivity measurement
  * slit lamp assessment and intra-ocular pressure measurement
  * ocular coherence tomography at the optic nerve head
  * visual field testing
  * OSOME (oxygen flow at the optic nerve head measurement)
  * Tropicamide
  Interventions: Procedure: Contrast sensitivity measurement; Procedure: Slit Lamp assessment and intra-ocular pressure measurement; Procedure: Visual field testing; Procedure: Oxygen flow at the optic nerve head measurement; Drug: Tropicamide; Device: OSOME
- CONTROL group (Historical database): * contrast sensitivity measurement
  * slit lamp assessment and intra-ocular pressure measurement
  * ocular coherence tomography at the optic nerve head
  * visual field testing
  * oxygen flow at the optic nerve head measurement (OSOME)
  * Under tropicamide
  Interventions: Procedure: Contrast sensitivity measurement; Procedure: Slit Lamp assessment and intra-ocular pressure measurement; Procedure: Visual field testing; Procedure: Oxygen flow at the optic nerve head measurement; Drug: Tropicamide; Device: OSOME

INTERVENTIONS:
Procedure: Contrast sensitivity measurement — Contrast sensitivity test is made with targets alternating black and white lines. The larger the lines are, easier it is to see them. Targets are distributed in 5 rows, each oriented at a different angle. Contrast sensitivity level is determined by the smallest target seen by the participant, line by line. This test is done under dim lightning with the habitual visual correction worn.
Procedure: Slit Lamp assessment and intra-ocular pressure measurement — Slit lamp is used to assess the presence of significant lens opacities known as Fabry cataracts. In fact, these opacities can induced a bias on the contrast sensitivity measurement and can increase the symptoms felt by the patient. A grade 2 (CFDI grading chart) of lens opacities is considered clinically significant and this will become an exclusion criteria for the following of the study. Intra-ocular pressure will be measured with a non contact tonometer (air pulsed) (Ocular Response Analyser, Reichert Instrumentation.)
Procedure: Visual field testing — Visual field will be assessed with an automated perimeter (Humphrey, Texas) using a threshold strategy. This implies that the subject has to identify not only if he perceives the visual stimulus but the minimal level of this stimulus (in decibels), to be seen, is also recorded. Visual field will be tested up to 30 degrees from the central point of fixation.
  In order to measure immediate variability of the visual testing among Fabry subjects, this test will be done at the beginning of the testing session (in the morning) and another time 1h00 later.
Procedure: Oxygen flow at the optic nerve head measurement — Pupils will be dilated with 1 drop of 1% tropicamide. The procedure is similar to the one used for taking a photo of the retina. Each measurement session represents a continuous recording of 20 simultaneous functions of reflectometry from the optic nerve area during 10 seconds.
  During all recording sessions, the systemic arterial oxygen saturation will be also monitored at the right index finger using a pulse oximeter (Escort M10, Invivo, Orlando, USA). Arterial blood pressure will be also monitored before and after the testing using a manual sphygmomanometer.
  Other Names: OSOME
Drug: Tropicamide — Used to dilate patient's pupil during testing
  Other Names: Mydriacyl® Mydriatic Tropicamide 1% Ophthalmic Drops; DIN 00001007
Device: OSOME — The OSOME system is the only technology able to perform on line and real time capillaries blood oxygenation measurement in the eye. The system operates with 1200 discreet wavelengths between 400 nm to 700 nm with 500 millisecond integration times. It is not invasive, functioning just like a fundus camera.
  Other Names: (O.S.O.M.E., US patent # 5,919,132;)

SUMMARY:
This study aimed to evaluate blood oxygenation at the optic nerve head in relation with visual field losses observed in many Fabry patients. Data collected allowed to evaluate if there is a link between these two entities.

Study lasted 2 years during which a limited number of Fabry patients had been compared to a control group to confirm any relationship between blood flow and field losses, and to see if these results varied over time.

HYPOTHESIS

1. Fabry patients will present significant differences in visual fields compared to control 2 There will be variability of the visual field defects on the long term but not on the short term 3 Blood oxygenation will be higher for Fabry patients 4 Blood volume at the optic nerve head will be the same for both groups.

DETAILED DESCRIPTION:
The first subjects who meet the following criteria will be enrolled in the study.

Inclusion criteria (Fabry group ):

* Aged over 18 years old
* Being diagnosed with Fabry disease

  * 3 subjects will be under enzyme replacement treatment for the treatment of Fabry disease.
  * 3 subjects will not receive enzyme replacement treatment
* Is fit to give legal consent.
* Is available for a period of 2 years

Inclusion criteria (CONTROL group ):

* Matched for age and sex with group A - 6 participants
* Being healthy, with no known chronic systemic disease nor acute disease at the moment of the recruitment
* Is fit to give legal consent.
* Is available for a period of 2 years

Exclusion criteria (Both groups):

* Presents with an active pathological ocular condition
* Presence of an abnormal optic nerve (congenital or acquired)
* Usage of topical ocular drug(s) at the time of selection
* To have known allergy to topical diagnostic drugs used in this study
* Usage of systemic medication with known effect on the visual field

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (Fabry group):

* Aged over 18 years old
* Being diagnosed with Fabry disease

  * 3 subjects will be under enzyme replacement treatment for the treatment of Fabry disease.
  * 3 subjects will not receive enzyme replacement treatment
* Is fit to give legal consent.
* Is available for a period of 2 years

Inclusion criteria (CONTROL group):

* Matched for age and sex with group A - 6 participants
* Being healthy, with no known chronic systemic disease nor acute disease at the moment of the recruitment
* Is fit to give legal consent.
* Is available for a period of 2 years

Exclusion Criteria:( both groups):

* Presents with an active pathological ocular condition
* Presence of an abnormal optic nerve (congenital or acquired)
* Usage of topical ocular drug(s) at the time of selection
* To have known allergy to topical diagnostic drugs used in this study
* Usage of systemic medication with known effect on the visual field

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients known as Fabry patients, already followed at Universite de Montréal eye clinic. COntrol will come from the normal clinical population seen at the same site.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Langis Michaud, OD M.Sc., Principal Investigator — Universite de Montreal
Locations (1):
- Universite de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pitz S, Grube-Einwald K, Renieri G, Reinke J. Subclinical optic neuropathy in Fabry disease. Ophthalmic Genet. 2009 Dec;30(4):165-71. doi: 10.3109/13816810903148004. PMID 19852573
- [Background] Kumagai K, Mitamura Y, Mizunoya S, Fujimoto N, Yamamoto S. A case of anterior ischemic optic neuropathy associated with Fabry's disease. Jpn J Ophthalmol. 2008 Sep-Oct;52(5):421-423. doi: 10.1007/s10384-008-0572-4. Epub 2008 Nov 11. No abstract available. PMID 18991052
- [Background] Feke GT, Riva CE. Laser Doppler measurements of blood velocity in human retinal vessels. J Opt Soc Am. 1978 Apr;68(4):526-31. doi: 10.1364/josa.68.000526. PMID 671138
- [Background] Diaconu V. Multichannel spectroreflectometry: a noninvasive method for assessment of on-line hemoglobin derivatives. Appl Opt. 2009 Apr 1;48(10):D52-61. doi: 10.1364/ao.48.000d52. PMID 19340124
- See also: web site of the School of Optometry University of Montreal — http://www.opto.umontreal.ca/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment group (Fabry) were actively recruited
Pre-assignment Details: Historic control group. Data collected from the files of patients - matched for age and sex- who consulted at Clinique Universitaire de la Vision. No active recruitment due to constraints in budget and manpower.
Groups:
- FABRY Group: * contrast sensitivity measurement
  * slit lamp assessment and intra-ocular pressure measurement
  * ocular coherence tomography at the optic nerve head
  * visual field testing
  * OSOME (oxygen flow at the optic nerve head measurement)
- CONTROL Group: * contrast sensitivity measurement
  * slit lamp assessment and intra-ocular pressure measurement
  * ocular coherence tomography at the optic nerve head
  * visual field testing
  * oxygen flow at the optic nerve head measurement (OSOME)
  C
Period: Overall Study
Arm/Group | FABRY Group | CONTROL Group
Started | 8 | 8 (Historical control group from database)
Completed | 6 | 8 (Historical control group from database)
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- CONTROL Group: * contrast sensitivity measurement
  * slit lamp assessment and intra-ocular pressure measurement
  * ocular coherence tomography at the optic nerve head
  * visual field testing
  * oxygen flow at the optic nerve head measurement (OSOME)
- Total: Total of all reporting groups
Arm/Group | FABRY Group | CONTROL Group | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants] — Population: The number analyzed in rows are detailled by category. The total of the participants in the 2 rows = overall number of participants. There is NO error
  Participants
    Hemizygotes- males: number analyzed (Participants) | 3 | 3 | 6
    Hemizygotes- males: <=18 years | 0 | 0 | 0
    Hemizygotes- males: Between 18 and 65 years | 3 | 3 | 6
    Hemizygotes- males: >=65 years | 0 | 0 | 0
    Heterozygotes- females: number analyzed (Participants) | 5 | 5 | 10
    Heterozygotes- females: <=18 years | 0 | 0 | 0
    Heterozygotes- females: Between 18 and 65 years | 4 | 4 | 8
    Heterozygotes- females: >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (14.8) | 43 (11.5) | 46 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygenation at the Optic Nerve Head
Description: OSOME measurement of the blood oxygenation at the optic nerve head
Time Frame: 2 years
Population: Fabry disease patients
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- Fabry: Fabry participants
- CONTROL Group: Historical control group Results extract from database
Arm/Group | Fabry | CONTROL Group
Number analyzed (Participants) | 8 | 8
percentage of oxygen saturation | 60.8 (5.4) | 65.3 (5.2)

2. Secondary Outcome: Field Defect
Description: Visual field defect using Frequency Doubling Technology (FDT)
  Results from FDT perimetry are reported using decibels of sensitivity. FDT perimetry has a manufacturer-provided internal normative database. (Deviation Plot). Results are compared to the normative database are shown on a gray scale plot based on probability levels. Screening tests preformed with the -5 screening test index ranges from P≥5% (worst) to P<1% (better)
  The global indices that are reported are the mean deviation (MD) and pattern standard deviation (PSD). MD values that fall below 5%, 2% 1% or 0.5 % normal probability levels are indicated with the appropriate label. Pattern Standard Deviation (PSD) represents how evenly the field loss is spread across the VF, thus indicative of localized loss. The PSD can only be equal to or greater than zero. The higher the PSD value, the greater the amount of irregularities with steeper slopes in the VF.
Time Frame: 2 years
Population: Fabry patients vs historic database
Measure: Mean (Standard Deviation); unit: Visual field Index (VFI)
Groups:
- FABRY: Threshold visual field VFI index
- CONTROL Group: Threshold visual field VFI index Historic database
Arm/Group | FABRY | CONTROL Group
Number analyzed (Participants) | 8 | 8
Visual field Index (VFI) | 98.4 (1.1) | 99.6 (0.6)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 years (Aug 2014- Sept 2016)
Description: There was no adverse event reported.
Groups:
- FABRY Group: * visual field testing
  * OSOME (oxygen flow at the optic nerve head measurement)
- CONTROL Group: * visual field testing
  * oxygen flow at the optic nerve head measurement (OSOME)
  C
Arm/Group | FABRY Group | CONTROL Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
The first obvious limitation is the nature of a pilot study, relying on a limited number of subjects. Sub-analysis is limited due to the fact that all except two Fabry participants have the same classic mutation (p.Ala348Pro), and all males and none women are on ERT. Consequently results analysis must be made with caution and can probably not be generalized to other Fabry's cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No